CLINICAL TRIAL: NCT03009630
Title: The Clinical Study of Electromagnetic Navigation Bronchoscopy (ENB) Guided Radiofrequency Ablation (RFA) for the Treatment of Early-stage Peripheral Lung Cancer
Brief Title: ENB Guided RFA for Early-stage Peripheral Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director, Endoscopy Department, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHCHE201604
Record Dates: First submitted 2016-12-30; First posted 2017-01-04 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Lung Cancer
Keywords: Electromagnetic navigation bronchoscopy(ENB); Radiofrequency ablation(RFA); Peripheral lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RFA group (Experimental): Patients with early-stage peripheral lung cancer will be performed RFA with the guidance of ENB. Post treatment response and follow up will be evaluated and carried out according to the standard procedure.
  Interventions: Procedure: RFA; Device: ENB

INTERVENTIONS:
Procedure: RFA — Patients diagnosed with early-stage NSCLC and signing the informed consent will be performed RFA under the guidance of ENB.
Device: ENB — ENB will be used to guide bronchoscope into the accurate location of the lesion during RFA.

SUMMARY:
The objective of the study was to evaluate the efficacy and safety of electromagnetic navigation bronchoscopy (ENB) guided radiofrequency ablation (RFA) for the treatment of early-stage peripheral lung cancer.

DETAILED DESCRIPTION:
The study is aimed to evaluate the efficacy and safety of ENB guided RFA for the treatment of patients with early-stage non-small cell lung cancer (NSCLC). The study is designed as a single-center prospective trial with one arm. The participating centers are Department of pulmonary medicine and endoscopy, Shanghai Chest Hospital affiliated to Shanghai Jiao Tong University, China. Patients diagnosed with early-stage NSCLC will be enrolled into the study. Fifty patients are expected to be enrolled totally.

ELIGIBILITY:
Inclusion Criteria:

1. Patients discovered with peripheral lung nodules that have demonstrated to be non-small cell lung cancer by pathology with the clinical stage of IA.
2. The tumors are solid or part-solid peripheral lung nodules and the length-diameter of the nodules are more than 10 mm and no more than 30 mm.
3. Patients are unsuitable for surgery assessed by multi-modality treatment and agree to the primary treatment of ablation.
4. Patients have good compliance and sign the informed consent.

Exclusion Criteria:

1. Patients cannot receive bronchoscopy for the severe cardiopulmonary dysfunction and other indications.
2. Patients have contraindications of general anesthesia.
3. Chest CT suggests that navigation bronchoscopy technology cannot guide treatment equipment to reach the peripheral lung lesion.
4. Chest CT or bronchoscopy shows that the bronchial lumen occlusion or deformation leading to the guided and treatment equipment cannot reach the peripheral lung lesion.
5. There are large blood vessels or important structures adjacent to peripheral lung lesion.
6. Researchers consider the patient do not fit for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Objective response rate（ORR）of participants as assessed by the modified RECIST criteria | Three months after ablation
  Objective response rate（ORR） is the proportion of patients with complete responses and partial responses according to the modified RECIST criteria.

SECONDARY OUTCOMES:
Progression-free survival (PFS) of participants | From the time of treatment to the time of disease progression or death with a follow-up period of 3 years
  Disease progression is evaluated by the variation of the tumor on computed tomography (CT) and/or positron emission tomography/computed tomography (PET/CT) according to modified RECIST criteria.
Overall survival（OS）of participants | From the time of treatment to the time of the patient death with a follow-up period of 5 years
  Overall survival（OS) is evaluated after the treatment of ablation until the patient death.

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From the time of treatment to one month after operation
  Complications refer to serious operation-related adverse events during and after the operation,such as pneumothorax, bleeding and infection.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, MD,PhD, Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harris K, Puchalski J, Sterman D. Recent Advances in Bronchoscopic Treatment of Peripheral Lung Cancers. Chest. 2017 Mar;151(3):674-685. doi: 10.1016/j.chest.2016.05.025. Epub 2016 Jun 10. PMID 27292045
- [Background] Koizumi T, Tsushima K, Tanabe T, Agatsuma T, Yokoyama T, Ito M, Kanda S, Kobayashi T, Yasuo M. Bronchoscopy-Guided Cooled Radiofrequency Ablation as a Novel Intervention Therapy for Peripheral Lung Cancer. Respiration. 2015;90(1):47-55. doi: 10.1159/000430825. Epub 2015 May 30. PMID 26044954
- [Background] Fernando HC, De Hoyos A, Landreneau RJ, Gilbert S, Gooding WE, Buenaventura PO, Christie NA, Belani C, Luketich JD. Radiofrequency ablation for the treatment of non-small cell lung cancer in marginal surgical candidates. J Thorac Cardiovasc Surg. 2005 Mar;129(3):639-44. doi: 10.1016/j.jtcvs.2004.10.019. PMID 15746749
- [Background] Dupuy DE, Fernando HC, Hillman S, Ng T, Tan AD, Sharma A, Rilling WS, Hong K, Putnam JB. Radiofrequency ablation of stage IA non-small cell lung cancer in medically inoperable patients: Results from the American College of Surgeons Oncology Group Z4033 (Alliance) trial. Cancer. 2015 Oct 1;121(19):3491-8. doi: 10.1002/cncr.29507. Epub 2015 Jun 19. PMID 26096694
- [Background] Anantham D, Feller-Kopman D, Shanmugham LN, Berman SM, DeCamp MM, Gangadharan SP, Eberhardt R, Herth F, Ernst A. Electromagnetic navigation bronchoscopy-guided fiducial placement for robotic stereotactic radiosurgery of lung tumors: a feasibility study. Chest. 2007 Sep;132(3):930-5. doi: 10.1378/chest.07-0522. Epub 2007 Jul 23. PMID 17646225
- [Background] Harms W, Krempien R, Grehn C, Hensley F, Debus J, Becker HD. Electromagnetically navigated brachytherapy as a new treatment option for peripheral pulmonary tumors. Strahlenther Onkol. 2006 Feb;182(2):108-11. doi: 10.1007/s00066-006-1503-2. PMID 16447018